CLINICAL TRIAL: NCT06249711
Title: Noninvasive Targeted Neuromodulation for Treatment of Food Addiction
Brief Title: Ultrasonic Treatment of Food Addiction
Acronym: USFADD
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Not activated at the site level
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Jan Kubanek, Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB_00175583
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-04

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active stimulation (Active Comparator): Low-intensity transcranial focused ultrasound stimulation of deep brain targets involved in food addiction
  Interventions: Device: Active stimulation with Diadem ultrasonic transducer array
- Sham stimulation (Sham Comparator): Zero-intensity transcranial focused ultrasound stimulation of deep brain targets involved in food addiction
  Interventions: Device: Sham stimulation with Diadem ultrasonic transducer array

INTERVENTIONS:
Device: Active stimulation with Diadem ultrasonic transducer array — Diadem ultrasonic transducer array delivers focused low-intensity ultrasound stimulation
  Arms: Active stimulation
Device: Sham stimulation with Diadem ultrasonic transducer array — Diadem ultrasonic transducer array delivers focused zero-intensity ultrasound stimulation
  Arms: Sham stimulation

SUMMARY:
This study will evaluate a new form of non-invasive deep brain therapy for food addiction. Low-intensity transcranial focused ultrasound stimulation will first be delivered using a range of stimulation parameters during psychophysical and physiological monitoring. A well-tolerated stimulation protocol will be selected for subsequent testing in a blinded randomized sham-controlled trial. The trial will evaluate brain target engagement using magnetic resonance imaging, Food Cravings Questionnaire-State, and changes in subject's weight over the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* History of at least one self-reported unsuccessful dietary effort to lose body weight
* Body mass index more than or equal to 30 kg/m^2 or more than or equal to 25 kg/m^2 with the presence of at least one of the following weight-related comorbidities: hypertension, dyslipidaemia, obstructive sleep apnoea, or cardiovascular disease.

Exclusion Criteria:

* Lifetime history of a serious suicide attempt
* MRI intolerance or contraindication
* Pregnant or breast feeding
* Diabetic (HbA1c more than 48 mmol/mol or 6.5%)
* A self-reported change in body weight more than 10 lbs within 60 days before screening
* Clinically inappropriate for participation in the study as determined by the study team

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03-03 (Actual); Primary Completion 2024-03-03 (Actual); Study Completion 2024-03-03 (Actual)

PRIMARY OUTCOMES:
Change in body weight (%) from baseline week 0 to week 16 | The body weight will be taken prior to each intervention (once per week)
  The body weight will be quantified with respect to baseline (100%), taken prior to the first intervention.
Number of participants who achieved body weight reduction >= 5% | Assessment at week 16
  Proportion of subjects who have lost at least 5% of their weight at week 16 relative to the baseline week 0.
Food Cravings Questionnaire-State | During and immediately after each weekly intervention
  This 15-item questionnaire measures immediate level of food craving, each item ranging from 1 (strongly disagree) to 5 (strongly agree). Higher total scores indicate stronger desire to eat.
Hamilton Depression Rating Scale, 17 item | For up to 16 weeks
  This 17-item questionnaire measures the severity of depression. Scores range between 0 (least severe) to 52 (most severe).

CONTACTS AND LOCATIONS:
Overall Officials: Jan Kubanek, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No